# Effect of Health Promotion on Allergic Rhinitis by Infrared-C Ray Irradiation

**Protocol ID: B10304016** 

Created Date: 6th August 2018

# **Participants:**

experimental group: 51 persons; control group: 51 persons

## **Inclusion criteria:**

- a. Adults that age 20 above and 50 below
- b. Clinical diagnosis confirmed as allergic rhinitis
- c. Conscious, no mental or cognitive impairment
- d. Able to read, write or communicate in Mandarin, Taiwanese or Hakka, and agreed to participate

# **Exclude criteria:**

- a. Inflammatory skin wounds on the back of the shoulder, neck or lower back
- b. Polyposis
- c. Acute and chronic sinusitis
- d. Vasomotor rhinitis

# **Experiment procedure:**



# **Experimental scheme:**



### **Assessment Scale:**

- 1. Basic demography questionnaire
- 2. Taiwanese Version of the 22-Item Sino-nasal Outcome Test (SNOT-20)
- 3. WHOQOL-BREF questionnaire (Allergic rhinitis questionnaire scale based on Taiwan's concise version of the World Health Organization Quality of Life Questionnaire)
- 4. Oral medication: type / dose / frequency /statistic in between

### **Examine:**

- 5. Ig-E blood examination (pre- and post-test)
- 6. Eosinophil cationic protein (pre- and post-test)

## **Method of Statistic:**

- 1. SPSS 18.0
- 2. The subjects were randomly grouped into experimental group and control group.
- 3. re-test was carried out before the experiment, 1<sup>st</sup> post-test was carried out at the 4<sup>th</sup> week and 2<sup>nd</sup> post-test was carried out at the 12<sup>th</sup> week. The data of the Pre- and post-test at the 4<sup>th</sup> & 12<sup>th</sup> week for both groups were statistically analyzed.
- 4. Independent t -test or chi-square test was carried out before the test for participant's basic information in both groups to examine the difference between the two groups.
- 5. Descriptive statistical analysis.
- 6. The data of pre- and post-test for two groups were compared by single-factor or two-factor analysis of variance (ANOVA).